CLINICAL TRIAL: NCT00099840
Title: Procalcitonin Guided Antibiotic Use in Acute Respiratory Tract Infections in Primary Care - A Randomized Controlled Trial
Brief Title: Procalcitonin Guided Antibiotic Use in Acute Respiratory Tract Infections (PARTI)-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Basel Institute of Clinical Epidemiology (BICE) (Other); Brahms AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PARTIS
Record Dates: First submitted 2004-12-21; First posted 2004-12-21 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2006-01

CONDITIONS: Respiratory Tract Infections
Keywords: common cold; pharyngitis; tonsillitis; rhinosinusitis; tracheo-bronchitis; otitis media; acute exacerbations of asthma; acute exacerbations of chronic pulmonary disease; community acquired pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Pharyngitis; Tonsillitis; Rhinosinusitis; Otitis Media; Community-Acquired Pneumonia

INTERVENTIONS:
Procedure: Procalcitonin guided antibiotic therapy

SUMMARY:
Acute respiratory tract infections (ARTI) are among the most frequent reasons for seeking medical attention in primary care. Although from predominantly viral origin, ARTIs are the most important condition for the prescription of antibiotics (AB), mainly due to the difficulty in primary care to differentiate between viral and bacterial etiology. Unnecessary AB use increases drug expenditures, side effects and AB resistance. A novel approach is to guide AB use by procalcitonin (ProCT), since serum levels are elevated in bacterial infections but remain lower in viral infections and inflammatory diseases.

We aim to compare a strategy based on evidence-based guidelines with ProCT guided AB therapy in ARTIs with respect to outcome (days with restriction) and AB use. Patients presenting with ARTIs to primary care physicians and are intended to be treated with AB based on guidelines will be included and randomized 1:1 either to standard management or to the ProCT guided prescription of AB. All participating physicians will receive evidence-based guidelines for the management of patients with ARTIs. Patients with ARTI and in need of ABs by physicians' clinical judgment and with informed consent will be randomized to ProCT plus guidelines ("ProCT group") versus only guidelines guided AB treatment ("control group"). In patients randomized to the ProCT group, the use of antibiotics will be more or less discouraged (<0.1 or <0.25 ug/L) or encouraged (>0.5 or >0.25 ug/L), respectively. A re-evaluation in patients with ProCT (<0.1 or <0.25 ug/L) after 6 to 24 hours is mandatory. All patients will be reassessed at day 3 and it is recommended to stop AB in the ProCT group as described above. Structured phone interviews at days 14 and 28 will be done in all patients from both groups.

DETAILED DESCRIPTION:
Background: Acute respiratory tract infections (ARTI) (i.e. common cold, pharyngitis, tonsillitis, rhinosinusitis, tracheo-bronchitis, otitis media, acute exacerbations of asthma (AEA) and of chronic pulmonary disease (AECOPD), and community acquired pneumonia (CAP)), are among the most frequent reasons for seeking medical attention in primary care. Although from predominantly viral origin, ARTIs are the most important condition for the prescription of antibiotics (AB), mainly due to the difficulty in primary care to differentiate between viral and bacterial etiology. Unnecessary AB use increases drug expenditures, side effects and AB resistance. A novel approach is to guide AB use by procalcitonin (ProCT), since serum levels are elevated in bacterial infections but remain lower in viral infections and inflammatory diseases.

Aim: To compare a strategy based on evidence-based guidelines with ProCT guided AB therapy in ARTIs with respect to outcome (days with restriction) and AB use.

Design: Randomized, controlled trial with an open intervention. Patients presenting with ARTIs to primary care physicians and are intended to be treated with AB based on guidelines will be included and randomized 1:1 either to standard management or to the ProCT guided prescription of AB.

Setting: Primary care providers in the Northwest of Switzerland from cantons with or without drug self dispensation (Basel-Stadt and Baselland).

Patients: 18 years or older, with ARTI of >1 and <28 days duration and in need of ABs based on the clinical judgment of the primary care physician. Excluded are patients without informed consent, not fluent in German, with AB pretreatment in previous 28 days or severe immune-suppression.

Endpoints: Primary: Days with restrictions from ARTI. Secondary: Rate of AB prescriptions, days with AB use, symptoms from ARTI, relapse rate from ARTI within 28 days, days with side effects from ABs and off work. Endpoints will be assessed at baseline, days 1 to 3 by the physicians. Structured phone interviews at days 14 and 28 will be done in all patients from both groups.

Intervention: All participating physicians will receive evidence-based guidelines for the management of patients with ARTIs. Patients with ARTI and in need of ABs by physicians' clinical judgment and with informed consent will be randomized to ProCT plus guidelines ("ProCT group") versus only guidelines guided AB treatment ("control group"). In patients randomized to the ProCT group the use of antibiotics will be more or less discouraged (<0.1 or <0.25 ug/L) or encouraged (>0.5 or >0.25 ug/L), respectively. A re-evaluation in patients with ProCT (<0.1 or <0.25 ug/L) after 6 to 24 hours is mandatory. All patients will be reassessed at day 3 and it is recommended to stop AB in the ProCT group as described above. Blood specimens for ProCT, taken from all patients, will be shipped by courier to the central lab and results will be reported within 2 hours.

Variables and measurement: Physicians have to consecutively enroll all patients with ARTI in whom they consider AB treatment. Baseline data on medical history and clinical items, additional diagnostic tests, co-morbidity and final prescribed treatment will be collected. The study will be conducted over a 12 month period in 2005.

Expected results: We assume noninferiority if at worst the new procedure leads to an increase on average of one day with restrictions compared to standard procedure with a reduced total AB use.

Our null hypothesis is: ProCT guided antibiotic management gives on average more than an extra day with restrictions than standard procedure.

Alternative hypothesis: ProCT guided antibiotic management gives on average at most one day with restrictions more than the standard procedure

Analyses: Analysis will be done based on the intention-to-treat principle. Sample size for type I error rate of 5% and type II error rate of 10% (i.e. 90% power) = 171. With allowance for a loss to followup of 10% the required sample size is 190 per treatment group. We intend to gain 24 primary care physicians to recruit the total of 380 patients.

Significance: Because of the high prevalence of ARTIs, this study will offer potential for improving the management of ARTIs in primary care by avoiding unnecessary ABs in patients with ARTIs, along with the prevention of AB resistance. For these reasons, it has high relevance for the Swiss health care system and for public health in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ARTI of >1 and <28 days duration
* In need of ABs based on the clinical judgment of the primary care physician

Exclusion Criteria:

* Patients without informed consent
* Not fluent in German
* AB pretreatment in previous 28 days
* Severe immune-suppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Days with restrictions from ARTI

SECONDARY OUTCOMES:
Rate of AB prescriptions
days with AB use
symptoms from ARTI
relapse rate from ARTI within 28 days
days with side effects from ABs and off work
cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Beat Muller, MD, Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, CH, Switzerland

REFERENCES:
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884